CLINICAL TRIAL: NCT03051568
Title: Evaluating Fluorine-18 Fluorodeoxyglucose Positron Emission Tomography /Computed Tomography With Liver SUVmax-based Criteria for Prognosis of Patients With Peripheral T-cell Lymphoma
Brief Title: Evaluating 18F-FDG PET/CT With Liver SUVmax-based Criteria for Prognosis of Patients With Peripheral T-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Xuejuan Wang,MD, Principal Investigator, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XW-PTCL-001
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: Lymphoma, T-Cell, Peripheral; Positron-Emission Tomography; Prognosis
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTCL patients with 18F-FDG PET/CT (Experimental): 18F-FDG PET/CT scans is to be evaluated using liver SUVmax-based criteria, Deauville 5-point criteria and reduction of SUVmax criteria
  Interventions: Device: 18F-FDG PET/CT

INTERVENTIONS:
Device: 18F-FDG PET/CT — 18F-FDG PET/CT will be conducted before, during and after chemotherapy. Patients were instructed to fast for at least 6 h before PET. The blood glucose level was measured to ensure that it was <200 mg/dL. 18F-FDG was intravenously administered at a dose of 3.7 MBq/kg. Approximately 60 ± 10 min post injection, a whole-body acquisition commenced in 6-8 bed positions (1 min/bed) using a hybrid system (PHILIPS Gemini TF) and covered from the base of the skull to the upper thigh, which was followed by CT in a non-contrast phase (modulated 100 mAs; 120 kV; slice thickness, 3 mm) for attenuation correction and anatomical localization purposes. The head acquisition was performed in one bed position (8-10 min/bed).

SUMMARY:
The purpose of this study is to evaluate whether a semi-quantitative interpretation using the liver SUVmax as reference can better interpret 18F-FDG PET/CT and predict disease progression during chemotherapy or survival in PTCL.

DETAILED DESCRIPTION:
In this study investigators develope a semi-quantitative interpretation using the liver SUVmax as reference to interpret 18F-FDG PET/CT. Positive lesions in PET were indicated as SUVmax of residues higher than the threshold or new 18F-FDG avid lesions. Investigators compare the prognostic accuracy of the liver SUVmax-based criteria with the 5-PS criteria and ΔSUVmax interpretation with respect to predicting disease progression during chemotherapy or survival in PTCL. Furthermore,investigators improve the prognostic ability of interim PET/CT by comparing the results to the clinical prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed PTCL
* treated using an anthracycline-containing regimen
* minimal follow-up at 6 months after the completion of first-line treatment
* complete medical history and clinicopathological data

Exclusion Criteria:

* secondary malignant disease
* serious infection or inflammation (e.g., HIV)
* primary central nervous system lymphoma
* hepatic or renal dysfunction.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in summed standardized uptake value (SUVmax) of lesion after 2 or 4 cycles | baseline(diagnosed by pathology and before chemotherapy) and 2 or 4 cycles after starting chemotherapy (each cycle 21days)

SECONDARY OUTCOMES:
3 year progression-free survival | up to 3 years after initial diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No